CLINICAL TRIAL: NCT03798652
Title: Improved Prediction of Functional Recovery After Revascularisation Using Combined Assessment of Myocardial Ischaemia and Viability by CMR - Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 247309
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2018-11

CONDITIONS: Cardiovascular Diseases; Ischemic Cardiomyopathy; Cardiac Ischemia
Keywords: Perfusion; Viability
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred for CABG: Patients with known coronary artery disease referred for isolated surgical revascularisation, who will be invited to attend our facility for a research CMR scan, a research 3D transthoracic echocardiogram and a 6 minute walk test
  Interventions: Device: Research CMR scan; Device: Research 3D transthoracic echocardiogram; Other: 6-minute walk test

INTERVENTIONS:
Device: Research CMR scan — CMR scanning at a 3Tesla scanner at King's College London
Device: Research 3D transthoracic echocardiogram — The scan is required to assess left ventricular systolic function
Other: 6-minute walk test — Sub maximal exercise that provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.

SUMMARY:
The study will investigate whether a new high resolution heart Magnetic Resonance Imaging scan, combining assessment of ischemia and viability by perfusion and Late Gadolinium Enhancement -Cardiac Magnetic Resonance is superior to Late Gadolinium Enhacement imaging alone in predicting functional recovery following revascularisation.

DETAILED DESCRIPTION:
Coronary artery disease, where the heart's blood supply is restricted by narrowings or blockages, is the commonest cause of heart failure. This condition is called ischaemic cardiomyopathy. In some patients, treating these narrowings/ blockages with by-pass surgery or stents, known as "revascularisation", helps improve the pumping strength of the heart but it is currently difficult to predict which patients will benefit. The best test the investigators currently have to predict who will benefit from revascularisation is an Magnetic Resonance Imaging scan of the heart which looks for how much the heart has been scarred. Hearts with no scar usually improve after revascularisation and hearts with lots of scar usually do not. However, lots of patients fall into the middle and have moderate amounts of scar. The Magnetic Resonance Imaging scan isn't good at predicting if this group of patients will benefit from revascularisation. Revascularisation procedures, including heart by-passes, are not without risk and often require time in intensive care, several days in hospital and a long recovery period at home. If the investigators can develop a better test which is more accurate at predicting whether hearts with moderate scar will improve then they will be able to provide better care for patients by ensuring only those patients who will get benefit from revascularisation are put through the procedure.

This study will investigate whether a new high-resolution heart Magnetic Resonance Imaging scan, which looks at not only levels of scar but also the quality of blood supply, is more accurate than current MRI scans at predicting heart recovery after revascularisation in patients with moderate amounts of scar.

ELIGIBILITY:
Inclusion Criteria:

1. Known coronary artery disease referred for isolated surgical revascularisation;
2. Wall motion abnormalities at rest in at least two adjacents segments on standard AHA model supplied by a diseased coronary artery;
3. LV EF <45%.

Exclusion Criteria:

1. Contraindications to CMR, adenosine and low-dose dobutamine;
2. GFR <30 ml/min
3. Decompensated heart failure requiring inotropic support, invasive or non-invasive ventilation or Intra-aortic Ballon Pump/left ventricular assist device therapy < 72 hours prior to enrolment;
4. Sustained Ventricular Tachycardia/Ventricular Fibrillation<72 hours prior to enrolment;
5. Implantable Cardioverter Defibrilator;
6. Pregnancy;
7. Age<18 years
8. Previous established diagnosis of non ischaemic cardiomyopathy;
9. Severe concomitant valvular disease;
10. Recente acute coronary syndrome(<4 weeks prior to enrolment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient will all the above inclusion criteria and none of the exclusion criteria will be identified from:
  * Referrals for cardiac MRI scans at King's College London;
  * Referrals for cardiac catheterisation at St. Thomas' Hospital;
  * Outpatient clinic referrals to St. Thomas's Hospital cardiovascular services;
  * Cardiovascular multi-disciolinary team meetings
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2019-03-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Recovery of the regional systolic function | 12 months
  Recovery will be defined as a reduction in average resting wall motion score equal or more than 1. The region of interest will be defined as the segments of myocardium subentended by the revascularised coronary stenosis.
  Segments will be considered to have been revascularised if surgical by-pass to the diseased coronary artery subtending the segment is considered successful by the surgical team at the time of surgery.

SECONDARY OUTCOMES:
Recovery of overall Left Ventricular ejection fraction | 12 months
Change in Left Ventricular end diastolic volume | 12 months

OTHER OUTCOMES:
Composite of all cause death hospitalisation for heart failure | 12 months
6- minute walk test | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Amedeo Chiribiri, Dr, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided